CLINICAL TRIAL: NCT06236932
Title: PRIN "SIDERALE": Susceptibility to Infectious Diseases in obEsity: an endocRine trAnslational socioLogic Evaluation
Brief Title: Susceptibility to Infectious Diseases in obEsity: an endocRine trAnslational socioLogic Evaluation, "SIDERALE"
Acronym: SIDERALE2020
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Roma La Sapienza (Other); University of Pisa (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); University of Rome Foro Italico (Other)
Responsible Party: Principal Investigator, Annamaria Colao, MD, PhD, Prof., Federico II University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIN SIDERALE
Record Dates: First submitted 2024-01-04; First posted 2024-02-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Type2diabetes; Lipodystrophy; Infections; Obesity Associated Disorder
Keywords: Obesity; Infections; Melatonin; Mediterranean Diet; Gut microbiota; Chronobiology
MeSH Terms: conditions — Obesity; Lipodystrophy; Infections | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mediterranean diet group (Active Comparator): At baseline (T0), all patients will be subjected to anthropometric determinations, including body weight and height for BMI calculation, body composition by mean of DXA Scan, blood, serum and urine collection, oral cavity swab and stool sampling. Patients will undergo a session of behavioural dietary counselling by which patients will be educated to adhere to a hypocaloric MD for the first 12w (T1).
  Interventions: Dietary Supplement: Mediterranean diet
- Mediterranean diet plus melatonin group (Active Comparator): After the first 12 w of the study (T2), all patients will continue a hypocaloric MD adding the supplementation with 1mg/die of melatonin before bedtime for other 12w.
  Interventions: Dietary Supplement: Mediterranean diet; Dietary Supplement: Melatonin supplementation

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — Hypocaloric Mediterranean Diet consist of a nutritional regimen with customized daily energy intake, calculated considering the Basal Metabolism and Physical Activity Level (LAF) of each patient. The distribution of macronutrients will be worked out as follows: ≃ 55-60% Carbohydrates (of which 80% are complex carbohydrates, pasta, bread, rice, whole grains and 20% simple sugars), ≃ 10-15% Proteins (of which the 60% of animal origin (meat, especially white) and 40% of vegetable origin (beans, chickpeas, lentils and legumes in general), ≃ 25-30% of lipids (predominantly olive oil).
Dietary Supplement: Melatonin supplementation — Melatonin (supplement formulation in capsules, 1mg/die one hour before sleep) will be associated with mediterranean diet for 12 w.
  Arms: Mediterranean diet plus melatonin group

SUMMARY:
Obesity is a life-threatening disease, defined by excessive fat accumulation that increases the risk of other diseases such as cardiovascular events, hypertension, diabetes and cancer. Obesity is also a risk factor for nosocomial infections and is associated with worse COVID-19 outcomes, although anthropometric measurements are not routinely recorded during hospitalization and lack of a registry data does not allow performing retrospective studies.Obesity is closely related to chronodisruption, characterized by deregulation of physiological and behavioral central and peripheral circadian rhythms contributing to the obesity-related metabolic impairment. Eating and sleeping time schedules are relevant synchronizers of humans' biological clock. Several studies suggest a role of dietary interventions in rewiring the circadian rhythm, with Mediterranean diet (MD) regulating nutritional patterns. Moreover, considering its positive impact on sleep quality, melatonin intake was suggested as a potential regulator of circadian rhythms. The relation between chronodisruption, obesity and infections has not been investigated, and a first proof of concept (Pilot study) will aim at investigating it. Three cohorts of obese patients with different aetiology (essential obesity, obesity with type 2 diabetes, genetic forms of obesity) and a cohort of lipodystrophic patients will be enrolled in the study, which is designed as a two-phases protocol. During the first phase (0-12 weeks (w)) patients will be subjected to dietary intervention with hypocaloric MD; in a second phase (12-24w), melatonin 1mg/die before sleep will be added to the hypocaloric MD. The susceptibility to infections will be investigated through the evaluation of 1) the number of events - i.e. flu- or flulike syndromes, skin, respiratory, digestive, urinary infections-per patient of the 4 groups and the blood assays to detect the infection with Epstein-Barr, Cytomegalovirus, Varicella, Measles and SARS-CoV-2 IgG and IgM; hepatitis C and hepatitis B core antibodies and Quantiferon TB Gold, 2) the clock genes rhythm and TLRs expression in patient immune cells at baseline, 12w and 24w.The mutual relationship between biomedical values, environmental and social conditions, and lifestyle habits will be evaluated by structured questionnaires. Validation of questionnaires to explore the susceptibility to infections is another delivery planned for the current study.

DETAILED DESCRIPTION:
The current project aims at investigating 1) the susceptibility to infectious disease in obese patients, the role of tailored dietetic schemes of Mediterranean diet (MD), and melatonin supplementation on infective events; 2) association of the oral and/or gut microbiota signature with bacterial or viral infections in the above described obese cohorts; 3) the mutual relationship between biomedical values, environmental conditions and lifestyle habits through structured questionnaires and therefore the possible impact of this study on the National Health System (NHS).

The role of melatonin as chronobiologic influencer of circadian metabolic processes and as anti-obesogenic and weight-reducing effector comes to the fore in these last decades. Moreover, melatonin is also known to possess anti-inflammatory and antioxidant properties that may ameliorate the condition of low-grade chronic inflammation (metaflammation) observed in patients with obesity. Nevertheless, although there has been a tremendous interest in the role of the clock genes in regulating metabolic processes, relatively less effort has been expended examining how the regulation of circadian rhythms and metabolic inputs can affect the susceptibility to infections. To address this question, Unit 1 will enroll patients with essential obesity (20 subjects, BMI :30-35 Kg/m2) and with genetic forms of obesity (20 subjects) of both genders, aged 18-65yrs, to the main proof of concept pilot study.

At baseline (T0), patients will be subjected to anthropometric determinations, including body weight and height for BMI calculation, body composition by mean of DXA Scan, blood, serum and urine collection, oral cavity swab and stool sampling. Patients will undergo a session of behavioural dietary counselling by which patients will be educated to adhere to a hypocaloric MD for the first 12w (T1) and to add to the MD the supplementation with 1mg/die of melatonin for other 12w (T2). The same patients will be visited and subjected to the anthropometric determinations and biological samples at T0, T1, T2 of protocol. The endpoints for Unit 1 will be: 1.to investigate the impact of tailored hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the number of events - i.e. flu- or flulike syndromes, skin, respiratory, digestive, urinary infections - per patient of the 4 groups, recording the number of infectious events during the clinical examinations in six months and 1 year follow up and detect the SARS-CoV-2, Epstein-Barr, Cytomegalovirus, Varicella and Measles IgG and IgM, hepatitis C and hepatitis B core antibodies and Quantiferon TB Gold (QFT-GIT). The obtained clinical results on infections events from the SIDERALE study will be used to formulate hypotheses for a prospective study and for the formulation of a specific validate questionnaire.

2.to assess the impact of a tailored hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on anthropometric determinations, glucose and lipid metabolism, thyroid and adrenal axis, leptin, adiponectin, IGFBP2, sirtuin 1 (SIRT1), ESR, high-sensitivity CRP, fibrinogen and inflammatory cytokines (TNF, IL-6, IL-1Beta, IL-18) and melatonin that will be evaluated at T0, T1, T2.

3.to assess the impact of a tailored hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the entrainment of circadian clock misalignment, evaluating clock gene expression by RT-qPCR in peripheral blood mononuclear cells (PBMC) and concomitantly, on the regulation of Toll like-receptors (TLRs) and suppressor cytokine signaling 3 (SOCS3), known to play a crucial role in eliciting immunity and improving the well-known susceptibility to infections in patients with obesity, all evaluated by RT-qPCR in PBMC of all patients cohorts at 8 am, 12 pm and 12 am.

4.to quantify the impact of our intervention on the NHS in terms of decrease of antibiotic and antiviral treatment and ER (emergency room) admissions in six months and 1 year of follow up.

Moreover, an in vitro analysis will be performed on 3T3-L1 cells (mouse pre-adipocytes). 3T3-L1 differentiated in adipocytes will be synchronized and treated with melatonin in presence of TLRs agonists (i.e.

lipopolysaccharide, Pam3CSK, ssRNA40, imiquimod). Evaluation of TLRs signalling pathway will be performed by western blot. Evaluation of inflammatory cytokines (TNF, IL-6, IL-1, IL-18) and chemokines (MCP-1, CXCL5) will be performed by CLIA and/or ELISA and/or western blot.

ELIGIBILITY:
Inclusion Criteria:

* essential obesity (BMI : 30-35 Kg/m2)
* genetic forms of obesity (BMI: 30-35 Kg/m2)
* obesity (BMI:30-35 Kg/m2) associated with T2DM
* obesity (BMI:30-35 Kg/m2) associated with endocrinopathies
* lipodystrophy

Exclusion Criteria:

* pregnancy, breast-feeding, alcohol and drug abuse, known severe haematological, cardiac, liver, kidney, mental diseases, hypogonadisms, hormonal treatments including estroprogestins, intolerance to melatonin or excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Investigation of the impact of hypocaloric MD and hypocaloric MD plus melatonin on the number of events - i.e. flu- or flulike syndromes, skin, respiratory, digestive, urinary infections in patients with obesity and lipodystrophy | Change from baseline at 3-6-12 months
  The primary outcome will be: to investigate the impact of tailored hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the number of events - i.e. flu- or flulike syndromes, skin, respiratory, digestive, urinary infections - per all patients, recording the number of infectious events,trough specific surveys, during the clinical and biochemical examinations in six months and 1 year follow up and detect the SARS-CoV-2, Epstein-Barr, Cytomegalovirus, Varicella and Measles IgG and IgM, hepatitis C and hepatitis B core antibodies and Quantiferon TB Gold (QFT-GIT).

SECONDARY OUTCOMES:
Change in body weight (kg) after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in body weight in all patients. Each determination will be assessed by scale and reported in kilograms (kg).
BMI modification after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy: body weight (kg) will be combined with height (m) to obtain BMI (kg/m^2) | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin will be evaluated by combining body weight (kg) with height (m) to calculate BMI (kg/m^2), where kg is a person's weight in kilograms and m2 is a person's height in metres squared.
Change in waist and hip circumference after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in waist and hip circumference, both reported in centimeters (cm).
Change in body composition assessed by Bioelectrical impedance analysis (BIA) after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy . | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on body composition will be assessed by Bioelectrical impedance analysis (BIA) in all patients.
Change in body composition assessed by DXA scan after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on body will be assessed by Dual-energy X-ray absorptiometry (DXA) scan.
Change in glucose profile assessed by blood glucose levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on glucose profile will be assessed in all patients by fasting blood glucose levels.
Change in glucose profile assessed by blood glycated hemoglobin (HbA1c) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on glucose profile will be assessed in all patients by fasting blood HbA1c levels.
Change in insulin profile assessed by blood insulin levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on insulin profile will be assessed in all patients by fasting blood insulin levels.
Change in insulin resistance assessed by homeostasis model assessment - insulin resistance (HOMA-IR) Index after hypocaloric MD and hypocaloric MD plus in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on insulin resistance will be assessed by HOMA-IR Index
Change in lipid profile assessed by blood total cholesterol levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on lipid profile will be assessed by fasting blood total cholesterol levels.
Change in lipid profile assessed by blood LDL cholesterol levels after hypocaloric MD and hypocaloric MD plus in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on lipid profile will be assessed by fasting blood LDL cholesterol levels
Change in lipid profile assessed by blood HDL cholesterol levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on lipid profile will be assessed by fasting blood HDL cholesterol levels in patients with obesity and lipodystrophy.
Change in lipid profile assessed by blood triglycerides levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on lipid profile will be assessed by fasting blood triglycerides levels.
Change in leptin levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in fasting blood leptin levels in all patients.
Change in adiponectin levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in fasting blood adiponectin levels in all patients.
Change in IGFBP2 (insulin like growth factor binding protein 2) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in fasting blood IGFBP2 levels in all patients.
Change in sirtuin 1 (SIRT1) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on variations in fasting blood sirtuin1 (SIRT1) levels in all patients.
Changes affecting the thyroid axis assessed by thyroid stimulating hormone (TSH) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on thyroid axis assessed by fasting blood thyroid stimulating hormone (TSH) levels in all patients
Changes affecting the thyroid axis assessed by free triiodothyronine (FT3) and free thyroxine (FT4) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on thyroid axis assessed by fasting blood free triiodothyronine (FT3) and free thyroxine (FT4) levels in all patients
Changes affecting the thyroid axis assessed by calcitonin levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on thyroid axis assessed by fasting blood calcitonin levels in all patients
Changes affecting the thyroid axis assessed by antibodies against thyroglobulin (AbTG) and against thyroperoxidase (AbTPO) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on thyroid axis assessed by fasting blood antibodies against thyroglobulin (AbTG) and against thyroperoxidase (AbTPO) levels in all patients
Changes in melatonin levels assessed by melatonin levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on melatonin levels assessed by fasting blood melatonin levels in all patients
Changes affecting the adrenal axis assessed by adrenocorticotropic hormone (ACTH) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on adrenal axis assessed by fasting blood adrenocorticotropic hormone (ACTH) levels in all patients
Changes affecting the adrenal axis assessed by cortisol levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on adrenal axis assessed by blood fasting cortisol levels in all patients
Changes affecting the adrenal axis assessed by dehydroepiandrosterone sulphate (DHEAS) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on adrenal axis assessed by blood fasting dehydroepiandrosterone sulphate (DHEAS) levels in all patients
Changes affecting the adrenal axis assessed by 17-hydroxyprogesterone (17-OHP) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on adrenal axis assessed by blood fasting 17-hydroxyprogesterone (17-OHP) levels in all patients
Change in low grade inflammation assessed by erythrocyte sedimentation rate (ESR) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on low grade inflammation assessed by blood ESR levels.
Change in low grade inflammation assessed by high-sensitivity CRP levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on low grade inflammation assessed by blood high-sensitivity CRP levels.
Change in low grade inflammation assessed by fibrinogen levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on low grade inflammation assessed by blood fibrinogen levels.
Change in low grade inflammation assessed by inflammatory cytokines (TNF, IL-6, IL-1Beta, IL-18) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on low grade inflammation assessed by blood inflammatory cytokines (TNF, IL-6, IL-1Beta, IL-18) levels. Evaluation will be performed by CLIA and/or ELISA and/or western blot.
Change in low grade inflammation assessed by inflammatory chemokines (MCP-1, CXCL5) levels after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin on low grade inflammation assessed by blood chemokines (MCP-1, CXCL5) levels. Evaluation will be performed by CLIA and/or ELISA and/or western blot.
Change in oral/gut microbiota after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months
  Assessment of the impact of hypocaloric MD and hypocaloric MD plus melatonin on oral/gut microbiota composition.
  Oral microbiota will be collected at fasting 8 am and at 4 pm. To study microbial communities associated to oral cavity, they will be sampled using swab while in order to study gut microbiota, stool will be collected. Samples will be stored at -80°C. From the two kinds of samples, DNA will be extracted and quantified using fluorimetric assay. Libraries of all the bacterial 16S DNA will be prepared using Microbiota solution A (V1-V2-V3 regions) for oral microbiome and Microbiota solution B (V3-V4-V6 regions) for gut microbiome.
Evaluation of hypocaloric MD and hypocaloric MD plus melatonin effects on circadian gene expression in peripheral blood mononuclear cells (PBMCs) in patients with obesity and lipodystrophy. | Change from baseline at 3-6 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the entrainment of circadian clock misalignment in patients with obesity and lipodystrophy will be assessed by evaluating clock gene expression through RT-qPCR in PBMCs at 8 am, 12 am and at 12 pm.
Evaluation of hypocaloric MD and hypocaloric MD plus melatonin effects on circadian Toll-like receptors (TLRs) gene expression in peripheral blood mononuclear cells (PBMCs) in patients with obesity and lipodystrophy | Change from baseline at 3-6 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the entrainment of circadian TLRs expression misalignment in patients with obesity and lipodystrophy will be assessed through RT-qPCR in PBMCs at 8 am, 12 am and at 12 pm.
Evaluation of hypocaloric MD and hypocaloric MD plus melatonin effects on circadian Suppressor Cytokine Signaling 3 (SOCS3) gene expression in peripheral blood mononuclear cells (PBMCs) in patients with obesity and lipodystrophy. | Change from baseline at 3-6 months
  The impact of hypocaloric MD and hypocaloric MD plus melatonin (supplement formulation, 1mg/die before sleep) on the entrainment of circadian SOCS3 misalignment in patients with obesity and lipodystrophy will be assessed through RT-qPCR in PBMCs at 8 am, 12 am and at 12 pm.
In vitro analysis conducted on 3T3-L1 cells (mouse pre-adipocytes) | Change from baseline at 3-6 months
  In vitro analysis will be performed on 3T3-L1 cells (mouse pre-adipocytes). 3T3-L1 cells differentiated into adipocytes will be synchronized and treated with melatonin to assess potential changes in clock gens and TLRs expression, evaluated by RT-qPCR. Moreover, adipocytes will be treated with melatonin in presence of TLRs agonists (i.e. lipopolysaccharide, Pam3CSK, ssRNA40, imiquimod) to assess potential modulation of TLRs signaling pathway evaluated by western blot.
Evaluation of adherence to MD (Mediterranean Diet) after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  Dietary habits will be assessed using a validated questionnaire (Predimed), based on the adherence to the Mediterranean Diet. This questionnaire generates a final score, determining whether patients are following the nutritional regimen correctly. Each question contributes 1 point, and the final score is categorized as follows: ≤5 indicates low adherence, 6 - 9 suggests medium adherence, and >10 reflects good adherence.
Evaluation of sleep habits after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  Sleep habits will be assessed using a validated questionnaire (Pittsburgh). This tool assesses perceived sleep quality through the evaluation of 19 items. The final score ranges from 0 to 21, where a score > 5 indicates poor sleep quality, while a score < 5 indicates good quality.
Evaluation of circadian rhythms after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  Circadian rhythms will be assessed using a validated questionnaire (Morningness - Eveningness Questionnaire MEQ-SA). This tool assesses morningness-eveningness in human circadian rhythms through 19 questions. The final score ranges from 16 to 86, where a score of 59 or more indicates an evening type, while a score of 41 or less indicates a morning type. Scores between 42 and 58 refers to intermediate types.
Reduction in the number of antibiotic and antiviral therapies after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  Assessment of the impact of our intervention on the NHS in terms of reduction in the number of antibiotic and antiviral therapies in all patients evaluated through patients' medical history
Reduction in the number of ER (emergency room) admissions for infections after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  Assessment of the impact of our intervention on the NHS in terms of reduction in the number of ER (emergency room) admissions for infections in all patients evaluated through patients' medical history
Assessment of social determinants' impact on susceptibility to infections after hypocaloric MD and hypocaloric MD plus melatonin in patients with obesity and lipodystrophy. | Change from baseline at 3-6-12 months.
  The assessment will be based on the administration of specific questionnaires and will include behavioral risk factor information, treatment compliance as well as techniques to reduce symptoms and features of obesity and lipodystrophy, overcome distress and improve coping, in order to promote a global improvement in quality of life. Power empowerment, self-efficacy and self-management will be investigated as intermediate outcomes to measure and report in terms of patient outcomes. Ultimate outcomes will include the individual's ability to obtain, process and understand basic health information needed to make appropriate health-related decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, Prof, Principal Investigator — Federico II University
Locations (4):
- Italy (4):
  - "Federico II" University of Naples, Department of Clinical and Molecular Endocrinology and Oncology, Naples
  - Università del Piemonte Orientale, Novara
  - University of Pisa, Pisa
  - "Sapienza" University of Rome, Roma

REFERENCES:
- [Background] Leitner DR, Fruhbeck G, Yumuk V, Schindler K, Micic D, Woodward E, Toplak H. Obesity and Type 2 Diabetes: Two Diseases with a Need for Combined Treatment Strategies - EASO Can Lead the Way. Obes Facts. 2017;10(5):483-492. doi: 10.1159/000480525. Epub 2017 Oct 12. PMID 29020674
- [Result] Barrea L, Muscogiuri G, Frias-Toral E, Laudisio D, Pugliese G, Castellucci B, Garcia-Velasquez E, Savastano S, Colao A. Nutrition and immune system: from the Mediterranean diet to dietary supplementary through the microbiota. Crit Rev Food Sci Nutr. 2021;61(18):3066-3090. doi: 10.1080/10408398.2020.1792826. Epub 2020 Jul 21. PMID 32691606
- [Result] Brown RJ, Araujo-Vilar D, Cheung PT, Dunger D, Garg A, Jack M, Mungai L, Oral EA, Patni N, Rother KI, von Schnurbein J, Sorkina E, Stanley T, Vigouroux C, Wabitsch M, Williams R, Yorifuji T. The Diagnosis and Management of Lipodystrophy Syndromes: A Multi-Society Practice Guideline. J Clin Endocrinol Metab. 2016 Dec;101(12):4500-4511. doi: 10.1210/jc.2016-2466. Epub 2016 Oct 6. PMID 27710244
- [Result] Ceccarini G, Pelosini C, Ferrari F, Magno S, Vitti J, Salvetti G, Moretto C, Marioni A, Buccianti P, Piaggi P, Maffei M, Santini F. Serum IGF-binding protein 2 (IGFBP-2) concentrations change early after gastric bypass bariatric surgery revealing a possible marker of leptin sensitivity in obese subjects. Endocrine. 2019 Jul;65(1):86-93. doi: 10.1007/s12020-019-01915-y. Epub 2019 Apr 3. PMID 30945111
- [Result] Chu Y, Yang J, Shi J, Zhang P, Wang X. Obesity is associated with increased severity of disease in COVID-19 pneumonia: a systematic review and meta-analysis. Eur J Med Res. 2020 Dec 2;25(1):64. doi: 10.1186/s40001-020-00464-9. PMID 33267871
- [Result] Pivonello C, Negri M, Patalano R, Amatrudo F, Monto T, Liccardi A, Graziadio C, Muscogiuri G, Pivonello R, Colao A. The role of melatonin in the molecular mechanisms underlying metaflammation and infections in obesity: A narrative review. Obes Rev. 2022 Mar;23(3):e13390. doi: 10.1111/obr.13390. Epub 2021 Dec 3. PMID 34861097
- [Result] Scheithauer TPM, Rampanelli E, Nieuwdorp M, Vallance BA, Verchere CB, van Raalte DH, Herrema H. Gut Microbiota as a Trigger for Metabolic Inflammation in Obesity and Type 2 Diabetes. Front Immunol. 2020 Oct 16;11:571731. doi: 10.3389/fimmu.2020.571731. eCollection 2020. PMID 33178196
- [Result] Turk Wensveen T, Gasparini D, Rahelic D, Wensveen FM. Type 2 diabetes and viral infection; cause and effect of disease. Diabetes Res Clin Pract. 2021 Feb;172:108637. doi: 10.1016/j.diabres.2020.108637. Epub 2021 Jan 13. PMID 33352263
- [Result] Watanabe M, Caruso D, Tuccinardi D, Risi R, Zerunian M, Polici M, Pucciarelli F, Tarallo M, Strigari L, Manfrini S, Mariani S, Basciani S, Lubrano C, Laghi A, Gnessi L. Visceral fat shows the strongest association with the need of intensive care in patients with COVID-19. Metabolism. 2020 Oct;111:154319. doi: 10.1016/j.metabol.2020.154319. Epub 2020 Jul 23. PMID 32712222
- [Result] Genoni G, Prodam F, Marolda A, Giglione E, Demarchi I, Bellone S, Bona G. Obesity and infection: two sides of one coin. Eur J Pediatr. 2014 Jan;173(1):25-32. doi: 10.1007/s00431-013-2178-1. Epub 2013 Oct 22. PMID 24146165